CLINICAL TRIAL: NCT04571398
Title: A Study of ApricityRx™ Digital Therapeutic for Management of Immune-Related Adverse Events in Patients on Immuno-Oncology Therapy
Brief Title: A Study of ApricityRx™ for Management of IR-AEs in Patients on Immuno-Oncology Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Apricity Health, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: AH0001
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Cancer
Keywords: cancer; immunotherapy; checkpoint inhibitors; immune-related adverse events
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ApricityRx mobile application — AE detection and monitoring software

SUMMARY:
Study of ApricityRx™ for Management of IR-AEs for patients on I-O therapy. Patients currently receiving immunotherapy will be asked to consent to participate in ApricityRx software platform mobile telephone application to report symptoms, view educational content in video form about IO and irAEs and communicate with site study team.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cancer diagnosis
* Prescribed treatment with immune-checkpoint inhibitor
* Age ≥ 18 years
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncomfortable with or unwilling to use digital or mobile technology
* Lack of a smart phone with compatible operating systems: iOS version 10 and above, or Android 6.0 Marshmallow
* Presence of any medical, psychological or social condition that, in the opinion of the investigator, would preclude participation in this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subject with a confirmed cancer diagnosis and prescribed checkpoint inhibitor therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate digital therapeutic mobile app to capture and transmit to care team patient-generated health data and access education content on IO and irAEs | 12 weeks
  Number of times and percentage of study participants who use the app to report patient reported health data during a 12 week period and access education videos.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Henick, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No